CLINICAL TRIAL: NCT04044027
Title: Evaluation of the Spark of Duval, an Innovative Teen Pregnancy Prevention Program
Brief Title: Evaluation of the Spark of Duval Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Svetlana Yampolskaya, Research Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00030249
Record Dates: First submitted 2019-07-17; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental)
  Interventions: Behavioral: S.P.A.R.K (Speaking to the Potential, Ability and Resilience inside Kids) Teen Pregnancy Prevention and Mentoring

INTERVENTIONS:
Behavioral: S.P.A.R.K (Speaking to the Potential, Ability and Resilience inside Kids) Teen Pregnancy Prevention and Mentoring — S.P.A.R.K is a curriculum-based group intervention for youth ages 11-17 living in out-of-home foster care. The curriculum consists of 23 topical lessons made up of a combination of educational and interactive activities on each topic. The curriculum covers four Adult Preparation Subjects (healthy relationships, educational and career success, healthy life skills, adolescent development) as well as mentoring, bully prevention, emotional competency, self-efficacy, communication, conflict resolution, and pregnancy prevention.
  Arms: Intervention Group

SUMMARY:
The S.P.A.R.K (Speaking to the Potential, Ability, and Resilience inside Kids) Teen Pregnancy Prevention and Mentoring program is being administered to youth (ages 11-17) living in out-of-home foster care in Duval County, Florida. Children's Home Society of Florida in Jacksonville received grant funding for the implementation and evaluation of the S.P.A.R.K program. The University of South Florida is examining the effects of intervention on reducing youth involvement in risky sexual behavior and incidents of teen pregnancy.

DETAILED DESCRIPTION:
The evaluation is conducting an individual randomized controlled trial to test the S.P.A.R.K. (Speaking to the Potential, Ability, and Resilience inside Kids) Teen Pregnancy Prevention and Mentoring intervention with youth assigned to either the intervention or control group. As youth are referred to the study, grantee staff confirm their eligibility and then work with the youth's child welfare case manager to obtain youth assent and parental consent. Once approximately 40 to 60 youth are recruited, grantee staff selects a day for baseline survey administration. Survey administration and group assignment take place at the grantee agency and incentives to complete the survey are provided including a gift card and snacks. All eligible youth with a signed assent and informed consent forms are invited to attend the baseline survey administration and group assignment. The evaluation team generates random numbers using computer software, and the grantee staff uses these numbers to indicate youth assignment to the intervention or control group, after youth have completed the baseline survey.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 11-17, living in out-of-home foster care in Duval County, FL (Florida) are eligible for participation. Only youth who have provided assent and have received parental/guardian informed consent are included in the study.

Exclusion Criteria:

* Youth who are teen parents, expectant parents, or currently living in residential facilities are excluded from the study.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in Sex Initiation | 3 months and 6 months
  Yes or No question regarding sexual activity
Change in Sexual Activity in the Past Three Months | 3 months and 6 months
  Number of times vaginal sex occurred in the past three months.
Change in Condom and Birth Control Use during Sex | 3 months and 6 months
  Frequency of condom use
Change in Pregnancy Occurrence | 3 months and 6 months
  Yes or No question regarding pregnancy
Change in Behaviors | 3 months and 6 months
  Survey questionnaire related to adolescent behaviors.

SECONDARY OUTCOMES:
Change in Connections with Peers | 3 months and 6 months
  Survey questionnaire related to connections with peers.
Change in Relationships with People | 3 months and 6 months
  Survey questionnaire related to relationships with people.
Change in Basic Life Skills | 3 months and 6 months
  Survey questionnaire related to basic life skills.
Change in Educational Expectations and Academic Success | 3 months and 6 months
  Survey questionnaire related to education expectations and academic successes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided